CLINICAL TRIAL: NCT02671422
Title: A Non-interventional Biomarker Study in Patients With Non-Small Cell Lung Cancer (NSCLC) of Adenocarcinoma Tumour Histology Eligible for Treatment With Vargatef® According to the Approved Label.
Brief Title: LUME BioNIS: a Biomarker Study in Patients With NSCLC
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199.223
Record Dates: First submitted 2016-01-29; First posted 2016-02-02 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — FPE tumour tissue and one blood sample. A buccal swab may replace the blood sample if not available.

SUMMARY:
At present there are no approved predictive tumour- or serum-derived biomarkers guiding usage of anti-angiogenic therapies in patients with adenocarcinoma of NSCLC.The objective of this NIS is to examine whether genetic/genomic markers (alone or combined with clinical covariates) could be used to predict OS in NSCLC patients eligible for treatment with Vargatef®. The investigations in this study are exploratory in nature and considered to be hypothesis generating. The results from these investigations may help to expand our understanding of the disease and the response to Vargatef®.

DETAILED DESCRIPTION:
Purpose:

ELIGIBILITY:
Inclusion criteria:

* Age = 18 years.
* Women and men with locally advanced, metastatic or locally recurrent NSCLC with histology of adenocarcinoma.
* Signed and dated written informed consent.
* Vargatef ® is initiated and administered in accordance with the SPC.
* Available fixed and paraffin embedded (FPE) tumour tissue routinely obtained at diagnosis and/or at re-biopsy before the initiation of the first line treatment (either block or slides, minimum of 10 slides and up to 20 slides if possible at 5µm thickness).

Exclusion criteria:

* Any contraindication to Vargatef® or docetaxel as specified in their respective labels.
* Vargatef® initiated more than 7 days prior to inclusion in this NIS.
* Patients participating simultaneously in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC patients under Vargatef® treatment according to label
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (71):
- Austria (2):
  - LK Krems, Krems
  - AKH - Medical University of Vienna, Vienna
- Belgium (7):
  - Brussels - UNIV Saint-Luc, Brussels
  - AZ Maria Middelares, Ghent
  - AZ Sint-Lucas - Campus Sint Lucas, Ghent
  - Ieper - HOSP Jan Yperman, Ieper
  - Liège - HOSP CHR de la Citadelle, Liège
  - Charleroi - UNIV CHU de Charleroi, Lodelinsart
  - Roeselare - HOSP AZ Delta, Roeselare
- Herlev and Gentofte Hospital, Herlev, Denmark
- Germany (10):
  - Gesundheit Nord gGmbH | Klinikverbund Bremen, Bremen
  - Florence-Nightingale-Krankenhaus der Kaiserswerther Diakonie, Düsseldorf
  - Pneumologisches Forschungsinstitut an der LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Onkologische Schwerpunktpraxis, Kaiserslautern
  - Klinik, Löwenstein, Löwenstein
  - Thoraxzentrum Bezirk Unterfranken, Münnerstadt
  - Klinikum Nürnberg, Nuremberg
  - Pius-Hospital, Oldenburg, Oldenburg
  - Caritas Klinik St. Theresia; Saarbrücken, Saarbrücken
  - SHG-Kliniken Völklingen, Völklingen
- Greece (3):
  - Athens Hospital of Chest Dis., Athens
  - University General Hospital of Heraklion, Heraklion
  - European Interbalkan Medical Centre, Thessaloniki
- Hungary (3):
  - National Koranyi TBC and Pulm. Internal Med. Clinic, Budapest
  - Lung Hospital of Matra, Dept. Pulmonology, Mátraháza
  - BAZ County Central Hospital and University Teaching Hospital, Miskolc
- Italy (2):
  - Azienda Ospedaliera Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia - Cervello, Palermo
- Lithuania (2):
  - Hospital of Lithuanian Univ.of HealthSciences Kauno Klinikos, Kaunas
  - National Cancer Institute, Vilnius, Vilnius
- Luxembourg - HOSP CH de Luxembourg, Luxembourg, Luxembourg
- Netherlands (7):
  - OLVG, locatie Oosterpark, Amsterdam
  - Ziekenhuis Gelderse Vallei, Ede
  - Martini Ziekenhuis, Groningen
  - Sint Jansdal Ziekenhuis, Harderwijk
  - Ziekenhuisgroep Twente locatie Hengelo, Hengelo
  - Tergooi Ziekenhuis, Hilversum
  - Maasstad Ziekenhuis, Rotterdam
- Spain (20):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario de Burgos, Buegos
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Complejo Hospitalario de Jaén, Jaén
  - Complejo Hospitalario Universitario Insular - Materno Infantil, Las Palmas de Gran Canaria
  - Hospital Severo Ochoa, Leganes - Madrid
  - Hospital de León, León
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Clínico San Carlos, Madrid
  - Hospital La Paz, Madrid
  - Hospital de Mataró, Mataró
  - Hospital Son Espases, Palma de Mallorca
  - Complejo Hospitalario de Navarra, Pamplona
  - CS Parc Taulí, Sabadell
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Virgen del Rocío, Seville
  - Hospital Virgen Macarena, Seville
  - Consorci Sanitari de Terrassa - Hospital de Terrassa, Terrassa
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
- Sweden (4):
  - Gävle Sjukhus, Gävle
  - Universitetssjukhuset, Linköping, Linköping
  - Karolinska Univ. sjukhuset, Stockholm
  - Akademiska sjukhuset, Uppsala
- United Kingdom (9):
  - Aberdeen Royal Infirmary, Aberdeen
  - Clatterbridge Cancer Centre, Bebington, Wirral
  - West Suffolk Hospital, Bury St Edmunds
  - Royal Devon and Exeter Hospital, Exeter
  - Ipswich Hospital, Ipswich
  - Airedale General Hospital, Keighley
  - James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle upon Tyne
  - Derriford Hospital, Plymouth

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-interventional study based on newly collected data in patients with Non-Small Cell Lung Cancer of adenocarcinoma tumour, who, for the first time, received Vargatef® as part of the routine treatment according to the approved label (new users design), to explore whether genetic or genomic markers could be used to predict Overall Survival.
Pre-assignment Details: Only subjects that met all the study inclusion criteria were to be entered in the study. All subjects were free to withdraw from the non-interventional study at any time for any reason given.
Groups:
- 200mg Vargatef®: Participants with Non-Small Cell Lung Cancer (NSCLC) were administered soft capsules of 200 milligram (mg) Vargatef® twice daily (except the day of docetaxel Infusion) in combination with 75mg/m² docetaxel every 21 days as indicated in the approved Labels of Vargatef® and docetaxel.
  Participants were followed-up every 6 months until they died, were lost to follow-up, withdrew consent, or until the required number of Overall Survival Events had occurred, whichever occurred first.
Period: Overall Study
Arm/Group | 200mg Vargatef®
Started | 260
Not Treated With Vargatef® | 3
Completed | 0
Not Completed | 260
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 68
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 7
Not completed — Progressive Disease | 156
Not completed — Worsening of Disease | 4
Not completed — Sponsor decision | 5
Not completed — Adverse Event unrelated to Vargatef® | 8
Not completed — Not treated with Vargatef® | 3
Not completed — Other not defined above | 3

BASELINE CHARACTERISTICS:
Population: Entered Set: All patients who entered the study, no matter if they acutally had taken Vargatef®.
Arm/Group | 200mg Vargatef®
Number analyzed (Participants) | 260
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 167
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52
  Not Hispanic or Latino | 208
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 256
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Survival (OS) Event
Description: Overall survival (OS) was defined as the time from start of entering the study to time of death. For the analysis of overall survival, participants were censored at the date of the last contact if the physician was no longer able to contact a participants or caregiver, and the vital status could not otherwise be determined. Enrolled participants who never received the combination therapy of docetaxel and Vargatef® were censored on the day of enrolment.
  Calculation of OS:
  For participants with known date of death: OS [days] = date of death - date of treatment start + 1 For participants known to be alive by the end of the study or at follow-up visit: OS (censored) [days] = date of last contact when the Patient was known to be alive - date of treatment start + 1.
Time Frame: From start of entering the study until death or last contact date, up to 42 months.
Population: Entered Set: All patients who entered the study, no matter if they actually had taken Vargatef®.
Measure: Count of Participants; unit: Participants
Arm/Group | 200mg Vargatef®
Number analyzed (Participants) | 260
Participants | 206
Statistical Analysis 1: Comparison: 200mg Vargatef®; Test type: Other; 1 year-survival rate = 0.342, 95% CI 2-sided [0.000 to 0.894] — Confidence interval is computed based on the LOGLOG method

ADVERSE EVENTS:
Time Frame: From first administration of study medication (Vargatef®) until 30 days after the last administration of study medication (Vargatef®), up to 807 days.
Description: For All-Cause Mortality the entered set (All patients who entered the study, no matter if they actually had taken Vargatef® ) was used.
  For serious and other adverse events, the Treated Set (All patients who were documented to have taken at least 1 Vargatef® dose) was used.
Arm/Group | 200mg Vargatef®
All-Cause Mortality (participants affected / at risk) | 209/260
Serious Adverse Events (participants affected / at risk) | 127/257
Other Adverse Events (participants affected / at risk) | 93/257
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 200mg Vargatef® (N=257)
Agranulocytosis (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 10
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Neutrophilia (Blood and lymphatic system disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 2
Vertigo (Ear and labyrinth disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 9
Enteritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Rectal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Chest pain (General disorders) | 1
Death (General disorders) | 1
General physical health deterioration (General disorders) | 1
Malaise (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Pain (General disorders) | 1
Performance status decreased (General disorders) | 3
Pyrexia (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 2
Campylobacter gastroenteritis (Infections and infestations) | 1
Clostridial infection (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Fournier's gangrene (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Meningoencephalitis herpetic (Infections and infestations) | 1
Neutropenic sepsis (Infections and infestations) | 2
Perirectal abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 13
Pulmonary sepsis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Septic shock (Infections and infestations) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
C-reactive protein increased (Investigations) | 2
White blood cell count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 66
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphasia (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Coma (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Device occlusion (Product Issues) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Embolism (Vascular disorders) | 1
Vena cava thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 200mg Vargatef® (N=257)
Diarrhoea (Gastrointestinal disorders) | 69
Nausea (Gastrointestinal disorders) | 24
Vomiting (Gastrointestinal disorders) | 15
Fatigue (General disorders) | 20
Decreased appetite (Metabolism and nutrition disorders) | 15

LIMITATIONS AND CAVEATS:
The planned number of 250 overall survival events could not be reached. Therefore, in agreement with the European Medicines Agency (EMA), the study was analysed earlier.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT02671422/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT02671422/SAP_001.pdf